CLINICAL TRIAL: NCT02122068
Title: Mentalizing Imagery Therapy for Major Depressive Disorder in Family Dementia Caregivers
Brief Title: Meditation for Dementia Caregivers Major Depressive Disorder in Family Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Friends of Semel Institute (Unknown); Morris A. Hazan Memorial Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMIT003
Record Dates: First submitted 2014-04-16; First posted 2014-04-24 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Mentalizing Imagery Therapy; Relaxation Recording
Keywords: Meditation; Mindfulness; Caregiver; Dementia; Depression
MeSH Terms: conditions — Dementia; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mentalizing Imagery Therapy (Experimental): Meditation and mindfulness 4 week program
  Interventions: Behavioral: Mentalizing Imagery Therapy
- Relaxation cd (Active Comparator): Listening to a relaxation cd
  Interventions: Behavioral: Relaxation cd

INTERVENTIONS:
Behavioral: Mentalizing Imagery Therapy — 4 week long meditation and mindfulness intervention
  Arms: Mentalizing Imagery Therapy
Behavioral: Relaxation cd
  Arms: Relaxation cd

SUMMARY:
Family dementia caregivers provide a needed service to relatives with dementia and to society, but are often at risk for consequences to their own health such as depression, reduced immune system function, and burnout. Mentalizing Imagery Therapy (MIT, previously known as Central Meditation and Imagery Therapy) is a novel group mindfulness and guided imagery intervention designed to help caregivers reduce depressive symptoms and cope with the stress of caregiving. We will conduct a pilot feasibility of MIT versus home relaxation practice with 24 dementia caregivers. Half of the caregivers will be randomly assigned to receive a relaxation recording, while the other half will receive MIT.

To measure the effects of MIT, we will obtain depression symptom ratings and questionnaires about psychological symptoms before and after MIT. We will also study the biological effects of MIT. We will do so by measuring brain activity, recording the pulse in order to determine variation in beat to beat intervals of the heart, and studying patterns of gene expression.

ELIGIBILITY:
Inclusion Criteria:

1. Caregivers of relatives with dementia who present to the UCLA Alzheimer and Dementia Care Program, or other UCLA geriatric or memory clinics for evaluation of dementia, cognitive impairment and/or co-existing behavioral disturbances.
2. Caregivers will be identified by the family member with dementia or the physician as the primary source of assistance and/or support
3. 45 years of age or older
4. Patient Health Questionnaire Score > 9
5. In contact with the individual with dementia at least three times/week for no less than one year, and a relative of the care-recipient (i.e., spouse or adult child).
6. Adequate written and oral fluency in English to understand and complete study forms and converse with study personnel.

Exclusion Criteria:

* Current diagnosis of schizophrenia or any psychotic disorder including psychotic depression, mania, alcohol or drug dependence, mental retardation, any pervasive developmental disorder or cognitive disorder (according to DSM-IV) criteria.

  2. Medically unstable, delirious, or terminally ill (e.g. medical illness requiring hospitalization or intense outpatient management, such as heart disease; heart attack in the past 6 months; congestive heart failure; severe heart arrythmias; unstable hypertension; poorly controlled diabetes; or pending surgery).

  3. Past history of skull fracture; cranial surgery entering the calvarium; space occupying intracranial lesion; stroke/ aneurysm; Parkinson's or Huntington's disease; or Multiple Sclerosis.

  4. Participants regularly practicing (≥ 2 times per week) any of the techniques utilized in the study to reduce stress: meditation, guided imagery, yoga.

  5. Active suicidal plan, or suicide attempt within the past month. 6. Excessive use of alcohol, i.e., men whose alcohol consumption exceeds 14 standard drinks per week or 4 drinks per day, and women whose alcohol consumption exceeds 7 standard drinks per week or 3 drinks per day.

  7. Needing to adjust or change anti-depressant treatment, including medications, psychotherapy, repetitive Transcranial Magnetic Stimulation (rTMS), Electroconvulsive Therapy (ECT), or Vagus Nerve Stimulation (VNS).

  8. Ideas of harm toward the care recipient, current violence, or an APS report on file.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 1 week post intervention (5 weeks)
  17 item rating scale, range of scores 0-52, higher scores indicate worse outcome

SECONDARY OUTCOMES:
Quick Inventory of Depression Symptoms - Self Report | 1 week post intervention (5 weeks)
  16 item rating scale, range of scores 0-27, higher scores indicate worse outcome

OTHER OUTCOMES:
State Trait Anxiety Inventory | 1 week post intervention (5 weeks)
  20 item rating scale, scores range from 20 to 80, higher scores indicate worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Felipe A Jain, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Jain FA, Nazarian N, Lavretsky H. Feasibility of central meditation and imagery therapy for dementia caregivers. Int J Geriatr Psychiatry. 2014 Aug;29(8):870-6. doi: 10.1002/gps.4076. Epub 2014 Jan 29. PMID 24477920